CLINICAL TRIAL: NCT06047873
Title: Clinical and Endoscopic Pattern in Children Presented With Upper and Lower Gastrointestinal Bleeding Insohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Bakhit Hussien, Resident-pediatric department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-23-07-18MS
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Upper and Lower Gastrointestinal Bleeding
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases (Experimental)
  Interventions: Device: Endoscopy

INTERVENTIONS:
Device: Endoscopy — clinical and endoscopic pattern in patients with upper and lower gastrointestinal bleeding

SUMMARY:
Gastrointestinal bleeding (GIB) is one of the most common conditions in the emergency department. Upper GIB is a major problem that has been decreasing over the past 20 years but still has high mortality rate. GIB usually manifests as hematemesis (vomiting of blood or coffee-ground-like material), melena (black or tarry stools), and hematochezia. UGIB appears as hematemesis in 40%-50%, and as melena or hematochezia in 90%-98%,However, patients with LGIB typically present with hematochezia, but right-sided colonic bleeding or small bowel bleeding may show as melena.

Endoscopy is the standard of care in the diagnosis and treatment of UGIB. It helps to identify the source of bleeding, establish the underlying etiology ,achieve hemostasis and provide prognostic information to predict the risk of rebleeding causes of UGIB are broadly divided into variceal and nonvariceal (peptic ulcer disease, reflux esophagitis, gastroduodenal erosions, tumors, vascular ectasia, etc. EGD is the diagnostic modality of choice for UGIB with more sophisticated investigations such as computed tomographic angiography and capsule endoscopy being rarely indicated where endoscopy is inconclusive .The primary diagnostic test for upper GI bleed workup is endoscopy. Sensitivity of 92 % - 98 % and specificity of 30 % - 100 % is present for endoscopy for the diagnosis of upper GI bleed. Severity scoring system like Rockall's score, helps to identify the patients who are at higher risk for rebleed and mortality.

Lower gastrointestinal ( GI ) haemorrhage is defined as bleeding distal to the ligament of Treitz. Most of the pathological lesions and haemorrhage in the lower GI tract are usually located in the rectum , sigmoid and left sided colon.It is usually suspected when patients complain of haematochezia (passage of frank bright red blood) or bloody diarrhea.Most of the bleeding from the lower GI tract stops spontaneously and patients usually have favorable outcomes compared to upper GI haemorrhage. However, morbidity and mortality tend to increase in older patients and with other pre existing co morbidities.

ELIGIBILITY:
Inclusion Criteria:

* children under 18years old who present with upper and lower gastrointestinal bleeding

Exclusion Criteria:

* bleeding due to systemic causes

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
endoscopy in upper and lower gastrointestinal bleeding and percentage of each disorder | 12 months
  detection of causes of gastrointestinal bleeding and percentage of each cause

IPD SHARING:
Plan to Share IPD: Undecided